CLINICAL TRIAL: NCT04781985
Title: Kafrelsheikh University Hospital
Brief Title: Prostatic Resection Cavity Stone Post Transurethral Resection of the Prostate (TURP). A Rare Case Scenario
Acronym: prostatic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Diaa Eldin Taha Ramadan Mohamed, lecturer of urology, Kafrelsheikh University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RS/20.12
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Prostate Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Cystoscopy

STUDY DESIGN:
Intervention Model Description: surgical treatment for bladder stone
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- suprapubic cystolithotomy (Experimental): Extraction of the vesical stone via open exploration of the bladder.
  Interventions: Procedure: cystoscopy

INTERVENTIONS:
Procedure: cystoscopy — extraction of the bladder stone via suprapubic incision
  Other Names: open cystolitholapaxy

SUMMARY:
Prostatic resection cavity stone post transurethral resection of the prostate (TURP). A rare case scenario

DETAILED DESCRIPTION:
Transurethral resection of the prostate (TURP) is the gold standard surgical therapy for lower urinary tract symptoms (LUTS) owing to senile prostatic enlargement. Following TURP, LUTS may persist in a percentage of patients. Persistent LUTS necessitates proper evaluation and management (1).

In a rare case report, delayed occurrence of storage and obstructive voiding symptoms after TURP can be caused by dystrophic calcification of the prostatic resection cavity and might be misinterpreted as post-TURP infection. The mechanism of dystrophic calcification entails minimizing tissue trauma by cautious removal of calcifications rather than performing extensive Re-TURP (2).

In our case, a rare presentation of storage LUTS as result of prostatic cavity stone extending into the bladder with same continuum, elicite the core issue of post TURP storage LUTS.

ELIGIBILITY:
Inclusion Criteria:

* patient with prostatic fossa stone post TURP

Exclusion Criteria:

* none

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
cystscopic evaluation of the prostate | one month
  evaluation of the prostatic fossa cavity post TURP
extraction of the bladder stone | one month
  surgical removal of the large bladder stone

CONTACTS AND LOCATIONS:
Locations (1):
- Diaa-Eldin Taha, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided